CLINICAL TRIAL: NCT06763575
Title: Efficacy of Surgical Glove-Compression Therapy As a Prevention of Paclitaxel-Induced Peripheral Neuropathy: Randomized Controlled Trial
Brief Title: Efficacy of Surgical Glove-Compression Therapy As a Prevention of Paclitaxel-Induced Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 67171
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Paclitaxel-induced Peripheral Neuropathy
Keywords: Paclitaxel; Surgical Glove-Compression Therapy; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: In the intervention group, patients wore double-layered surgical gloves, one size smaller than measured, covered by large cotton gloves on both hands, for 30 minutes before, during, and after chemotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical Glove-Compression Therapy (Experimental): Patients wore double-layered surgical gloves, one size smaller than measured, covered by large cotton gloves on both hands, for 30 minutes before, during, and after chemotherapy.
  Interventions: Device: Surgical Glove-Compression Therapy
- non-compressive plastic gloves (Placebo Comparator): Patients wore non-compressive plastic gloves, covered by large cotton gloves on both hands, for 30 minutes before, during, and after chemotherapy.
  Interventions: Device: non-compressive plastic gloves

INTERVENTIONS:
Device: Surgical Glove-Compression Therapy — In the intervention group, patients wore double-layered surgical gloves, one size smaller than measured, covered by large cotton gloves on both hands, for 30 minutes before, during, and after chemotherapy.
  Arms: Surgical Glove-Compression Therapy
Device: non-compressive plastic gloves — In the control group, patients wore non-compressive plastic gloves, covered by large cotton gloves on both hands, for 30 minutes before, during, and after chemotherapy.
  Arms: non-compressive plastic gloves

SUMMARY:
The aim of this randomized controlled trial (RCT) is to compare the incidence of paclitaxel-induced grade 2 or higher sensory peripheral neuropathy, evaluated using the CTCAE version 5.0, between patients receiving surgical glove-compression therapy (SGCT) and those in the control group.

The main question is whether SGCT is effective in preventing paclitaxel-induced sensory peripheral neuropathy.

* Intervention group: receive SGCT.
* Control group: receive non-compressive plastic gloves.

DETAILED DESCRIPTION:
1. The study aims to test the hypothesis that SGCT is effective in preventing paclitaxel-induced peripheral neuropathy.
2. The primary objective is to determine the incidence of grade 2 or higher paclitaxel-induced sensory peripheral neuropathy, assessed using the CTCAE version 5.0. Secondary objectives include evaluating the incidence of grade 2 or higher paclitaxel-induced motor peripheral neuropathy using CTCAE version 5.0, the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) score, the incidence of grade D or higher paclitaxel-induced sensory and motor peripheral neuropathy as measured by the Patient Neurotoxicity Questionnaire (PNQ), and the outcomes from the monofilament test.
3. Sample size formula based on Bernard R. Fundamentals of biostatistics. 5th ed. Duxbery: Thomson learning; 2000. Enrollment of 36 patients.
4. Randomization into two groups. The intervention arm will receive SGCT, while the control arm will receive non-compressive plastic gloves. The duration of treatment is 9 weeks.
5. Enrollment and data monitoring are assessed by staff at the Oncology Unit, Rajavithi Hospital, and the data will be recorded in a computer-based information system.
6. Data assessment will be conducted on weeks 0, 3, 6, and 9 during the chemotherapy treatment.
7. Data analyzed by descriptive and inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age 18 years or older at the time of signing Informed Consent Form
* Patients with any pathological diagnosis of solid tumor, such as breast cancer or lung cancer
* Patients scheduled to be receiving intravenous paclitaxel or paclitaxel-based regimen every 3 weeks

Exclusion Criteria:

* Patients whose received chemotherapeutic agents that could cause neuropathy, e.g. taxane-based or platinum-based chemotherapy and anti-microtubule
* History of neuropathy
* History of carpal tunnel syndrome
* History of allergic reactions to latex or gloves
* Patients receiving treatments that may treat neuropathy, e.g. amitriptyline, gabapentin, Acetyl L-Carnitine and Ganglioside-monosialic acid, acupuncture, cryotherapy or exercise therapy
* History of Raynaud phenomenon
* History of wounds or large scars on hands
* Pregnancy or breastfeeding
* History of poorly controlled diabetes; HbA1c>6.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher paclitaxel-induced sensory peripheral neuropathy using CTCAE version 5.0. | 9 weeks
  The incidence of grade 2 or higher paclitaxel-induced sensory peripheral neuropathy was evaluated using the CTCAE version 5.0 for both the intervention and control groups.

SECONDARY OUTCOMES:
Incidence of grade 2 or higher paclitaxel-induced motor peripheral neuropathy using CTCAE versions 5.0 | 9 weeks
  The incidence of grade 2 or higher paclitaxel-induced motor peripheral neuropathy was evaluated using the CTCAE version 5.0 in both the intervention and the control groups.
FACT/GOG-NTX scores | 9 weeks
  FACT/GOG-NTX scores in both the intervention and the control group.
Incidence of grade D or higher paclitaxel-induced sensory and motor peripheral neuropathy using the PNQ | 9 weeks
  The incidence of grade D or higher paclitaxel-induced sensory and motor peripheral neuropathy using the PNQ in both the intervention and the control group.
Monofilament test results | 9 weeks
  Monofilament test results in both the intervention and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sunatee Sa-nguansai, M.D., Study Director — Department of Medical Services Ministry of Public Health of Thailand; Saowani Thantaviraya, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand; Kunlatida Maneenil, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand; Piyawan Tienchaiananda, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand; Songwit Payapwattanawong, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Medical Oncology Unit, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2024 - December 2025